CLINICAL TRIAL: NCT02216318
Title: A Study of Two Different Light Conditions for Healthy Subjects Above 65 Years
Brief Title: Energy-efficient and Health Promoting Light for Elderly People
Acronym: light-age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Elforsk (Unknown); Albertslund Kommune (Unknown); Gate 21 (Unknown); DTU Fotonik (Unknown); VISO systems (Unknown); AF Lightning (Unknown); Philips Healthcare (Industry); Statens Byggeforskningsinstitut (Unknown)
Responsible Party: Principal Investigator, Line Kessel, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-3-2013-085
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Sleep
Keywords: sleep; circadian; melatonine; pupil response
MeSH Terms: interventions — Blue Light

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- red light (Placebo Comparator): red light during the whole day
  Interventions: Other: blue light
- Blue light (Active Comparator): Blue light during early day
  Interventions: Other: blue light

INTERVENTIONS:
Other: blue light

SUMMARY:
to investigate the effect of two lightning conditions on sleep hypothesizing that sleep length is influenced by the color of light during daytime

DETAILED DESCRIPTION:
Lightning conditions seems to be important for the length and quality of sleep, as light have an influence on the production of the sleep hormone (melatonin) and the the circadian rhythm. Entrainment of the circadian rhythm to the surroundings is accomplished by light-sensitive retinal ganglion cells and these cells are sensitive to blue light.

Based on previous research, blue light early in the day and abscence of blue light during evening is important for the entrainment.

In this study, lightning conditions in the home of healthy subjects are set to either blue enriched or red enriched from 8 a.m to 1. p.m. The lightning condition is based on a randomization protocol in a cross-over study for 3 weeks in each condition, separated by a one week pause.

ELIGIBILITY:
Inclusion Criteria:

* age 65 to 85 years

Exclusion Criteria:

* Conditions which will interfere by the primary endpoint as evaluated by the medical doctor

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Sleep length | 1 week
  The mean of sleep length during the last week of each light period

SECONDARY OUTCOMES:
actigraphy | 1 week
  mean sleep efficiency during the last week in each light period

OTHER OUTCOMES:
pupillometry | the last day of each light period
  the pupillary response to blue and red light
melatonin | the last day of each light period
  timing of melatonin onset
Questionnaire | 3 weeks
  Questionnaire count

CONTACTS AND LOCATIONS:
Overall Officials: Line Kessel, MD, Principal Investigator — Glostrup University Hospital, Copenhagen